CLINICAL TRIAL: NCT04877093
Title: Repurposing Low-Dose Clonidine for PTSD in Veterans
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00105944; 20-1057 (Other: Advocate Aurora Health Care)
Record Dates: First submitted 2021-01-28; First posted 2021-05-07 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: PTSD; Posttraumatic Stress Disorder; Sleep
Keywords: PTSD; veterans; military; sleep; adrenergic receptor
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Clonidine

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, blinded crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacist will determine the groups for each patient and will not reveal groups to anyone on the study team or the participant until they have finished the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Clonidine Phase (Experimental): Participants will receive clonidine titrations across 6 weeks. Note that this is a crossover design, so patients will move across phases.
  Interventions: Drug: Clonidine Pill
- Placebo Phase (Placebo Comparator): Participants will receive placebo titrations across 6 weeks. Note that this is a crossover design, so patients will move across phases.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Clonidine Pill — The study will use a flexible-dose adjustment schedule to identify the minimum dose needed to alleviate symptoms while also ensuring acceptable adverse effects. In other words, all subjects will start at the minimum dose (0.1 mg/night). Near the end of every week, each subject will be assessed for symptom alleviation and adverse events by asking the patient two questions from the CAPS-5 (questions B2 and E6. At baseline, each patient will have scored a ≥3 on each of these questions. If one or both scores remain at ≥3 and if any reported adverse events are marked acceptable by both the clinician and subject, then the dosage for the following week will be increased one level according to the titration chart. However, if both scores for these questions are ≤2 and any current adverse events are acceptable, then the dosage will remain the same. Finally, if any adverse events are deemed unacceptable, the clonidine dosage will be reduced to the lowest acceptable daily dosage.
  Arms: Clonidine Phase
Other: Placebo — Blinded placebo capsules will be provided to participants.
  Arms: Placebo Phase

SUMMARY:
Hypothesis: Veterans with PTSD prescribed clonidine will demonstrate improvements in PTSD symptoms, including daytime, nighttime, and sleep-related behaviors.

DETAILED DESCRIPTION:
Military veterans with Posttraumatic Stress Disorder (PTSD) suffer emotionally, physically, and socially. They have higher rates of suicide,1 issues with anger/aggression,2 substance use disorder,3 or other life difficulties (e.g., mental health disorders, marriage instability, unemployment).4 However, current first-line treatments are only effective for around half of patients receiving treatment.5,6 This is problematic given that PTSD is relatively common with a lifetime prevalence in US veterans of 10 - 31%3,7 meaning that many military veterans and their families are suffering for lack of effective treatments.

PTSD symptoms can be categorized into four clusters: re-experiencing, avoidance, cognitive or mood disturbances, and hyperarousal/reactivity.8 Symptoms may occur during the day or at night, thus disrupting sleep. Many symptoms are thought to be mediated through noradrenergic pathways. Specifically, noradrenergic overactivity may directly or indirectly affect irritability/aggression, hypervigilance, ability to concentrate, startle reactions, and sleep or other nighttime symptoms.9 These nighttime disruptions are especially problematic given that lack of sleep can exacerbate other PTSD symptoms directly or through associations with increased depression, heightened anxiety, and unstable mood/affect.10-12 Selective serotonin reuptake inhibitors (SSRI) are a first-line pharmacotherapy for PTSD, yet SSRIs do not target noradrenergic pathways, have reduced efficacy in veterans,13 and only weakly impact nighttime symptoms.11,14,15

To directly address hyperarousal and sleep, previous studies have tested medications targeting the noradrenergic pathway or sleep interventions, resulting in promising outcomes for a subpopulation of veterans with PTSD.16-27 Studies on prazosin, an antagonist of post-synaptic α1 noradrenergic receptors, have shown promise for veterans with PTSD.16,18 Clonidine is similar to prazosin and is proposed to have similar effects on PTSD; however, whereas prazosin and blocks the effects of norepinephrine, clonidine decreases norepinephrine release 28 and could therefore have greater effects on hyperarousal. Retrospective, open-label studies have suggested that clonidine use is associated with improvement in PTSD.16,17 However, no prospective studies have been published testing the effects of clonidine on PTSD, either in veterans or any other population.

Hypothesis: Veterans prescribed clonidine will demonstrate improvements in PTSD symptoms, including daytime, nighttime, and sleep-related behaviors.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* US military veteran
* Currently has PTSD diagnosis as determined by clinical diagnosing or by the PI
* Screening score on PCL5 minimum of 40 (per data from previous studies36-38, a PCL5 score of 40 is roughly equivalent to a CAPS score of 30)
* Scores ≥10 on PCL5 items 1-5 (intrusion) or scores ≥10 on PCL5 items 15-20
* From PCL5 questionnaire, must score the following minimum in each of the following categories:

  * 1x score of 2 on Questions 1-5
  * 1x score of 2 on Questions 6-7
  * 2x score of 2 on Questions 8-14
  * 2x score of 2 on Questions 15-20
* Has score ≥3 on CAPS nightmare items B2 and E6
* Speaks and understands English
* Willing to come into the clinic as programmed

Exclusion Criteria:

* Pregnant or breastfeeding
* At Moderate or High risk of suicide based on "past month" column of the Columbia-Suicide Severity Rating Scale (CSSR-S) screen version - recent.
* Has acute or unstable mental illness or any cognitive issues which the PI determines would interfere with engagement in the study (e.g., active schizophrenia, uncontrolled bipolar, history of neurocognitive impairment, history of moderate-severe traumatic brain injury)
* Currently receiving exposure therapy
* Recently enrolled (<1 month) in other behavioral health therapies (exclusions made at the PI's discretion depending on therapy type and length since admission)
* Urgent hypertension (BP above 160/100) or symptomatic of hypertension (having a hypertensive emergency)
* Blood pressure under 100/60 or symptoms of low blood pressure (light headedness, dizziness, heart palpitations, or other symptoms as determined by clinician).
* Any contraindications to taking clonidine such as:

  * Known hypersensitivity to clonidine
  * History of 2nd or 3rd degree atrioventricular block
  * History of sinus bradycardia
  * History of pheochromocytoma
  * History of Raynaud's phenomenon
  * Stage 5 Kidney disease
  * Recent myocardial infarction (<6 months)
  * History of cerebrovascular disease or recent stoke (<6 months)
* Have used any of the following drugs in the past 30 days, unprescribed or not used as prescribed:

  * Heroin
  * Other opiates/analgesics
  * Barbiturates
  * Other sedatives/, hypnotics, or tranquilizers
  * Cocaine
  * Amphetamines
  * Cannabis
  * Hallucinogens
  * Inhalants
* Currently have any of the following diagnoses:

  * Opioid use disorder
  * Cocaine use disorder
  * Alcohol use disorder
  * Cannabis use disorder
  * Sleep apnea diagnosis with verbal indication of non-adherence to treatment
* Were prescribed clonidine within the last 6 months

  * Any α2 agonist

    * Catapres/Kapvay (clonidine)
    * Aldomet (Methyldopa)
    * Zanaflex (Tizanidine)
    * Intuniv (Guanfacine)
    * Lucemyra (Lofexidine)
  * Any α1-adrenergic antagonist

    * Prazosin
    * Terazosin
    * Doxazosin
    * Silodosin
    * Alfuzosin
    * Tamsulosin
  * Any opiate (e.g., buprenorphine, hydrocodone, oxycodone)
  * Any antipsychotic medication

    * Haldol (haloperidol)
    * Loxitane (loxapine)
    * Mellaril (thioridazine)
    * Moban (molindone)
    * Navane (thiothixene)
    * Prolixin (fluphenazine)
    * Serentil (mesoridazine)
    * Stelazine (trifluoperazine)
    * Trilafon (perphenazine)
    * Thorazine (chlorpromazine)
    * Abilify (aripiprazole)
    * Clozaril (clozapine)
    * Geodon (ziprasidone)
    * Risperdal (risperidone)
    * Seroquel (quetiapine)
    * Zyprexa (olanzapine)
  * Benzodiazepines
  * Cyproheptadine
* Based on PI or study team assessment is cognitively unable to engage in the study
* Has a legal guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pittsburgh Sleep Quality Index (PSQI) at 6 weeks into phase | Week 6 of Current Phase
  Scored 0-21, where higher scores indicate worse sleep quality.
Change from Baseline in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) questions B2 and E6 at 6 weeks into phase | Week 6 of Current Phase
  Measures PTSD symptoms on sleep, with each question scored 1-4, where higher scores indicate more severe symptoms.
Change from Baseline in PTSD Checklist-Military Version (PCL-5) at 6 weeks into phase | Week 6 of Current Phase
  Includes 20 items with a severity score range 0-80. Includes the ability to treat each item rated as 2 = "Moderately" or higher as a symptom endorsed, which allows following the DSM-5 diagnostic rule which requires at least: 1 Criterion B item (questions 1-5), 1 Criterion C item (questions 6-7), 2 Criterion D items (questions 8-14), 2 Criterion E items (questions 15-20). In general, use of a cutoff score tends to produce more reliable results than the DSM-5 diagnostic rule.

SECONDARY OUTCOMES:
Change from Baseline in Patient Health Questionnaire (PHQ9) at 6 weeks into phase | Week 6 of Current Phase
  Scored 0-27, where higher scores indicate greater depression
Change from Baseline in Sleep Diary at 6 weeks into phase | Week 6 of Current Phase
  Qualitative differences in the sleep diary responses
Change from Baseline in quality of life scale (Q-LES-Q-SF) at 6 weeks into phase | Week 6 of Current Phase
  Scored 16-80, where higher scores indicate greater quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Burek, MD, MS, Principal Investigator — Wake Forest University Health Sciences; Michael Fendrich, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora Psychiatric Hospital, Wauwatosa, Wisconsin, United States

REFERENCES:
- [Background] Kang HK, Bullman TA. Risk of suicide among US veterans after returning from the Iraq or Afghanistan war zones. JAMA. 2008 Aug 13;300(6):652-3. doi: 10.1001/jama.300.6.652. No abstract available. PMID 18698062
- [Background] Buchholz KR, Bohnert KM, Sripada RK, Rauch SA, Epstein-Ngo QM, Chermack ST. Associations between PTSD and intimate partner and non-partner aggression among substance using veterans in specialty mental health. Addict Behav. 2017 Jan;64:194-199. doi: 10.1016/j.addbeh.2016.08.039. Epub 2016 Aug 31. PMID 27636157
- [Background] Norman SB, Haller M, Hamblen JL, Southwick SM, Pietrzak RH. The burden of co-occurring alcohol use disorder and PTSD in U.S. Military veterans: Comorbidities, functioning, and suicidality. Psychol Addict Behav. 2018 Mar;32(2):224-229. doi: 10.1037/adb0000348. PMID 29553778